CLINICAL TRIAL: NCT06643572
Title: Comparing the Effectiveness of Using Patient Imaging and Virtual Reality-based Simulation Prior to Challenging Lumbar Transforaminal Epidural Steroid Injections: a Randomized Controlled Trial
Brief Title: Comparing of Using Patient Imaging and Virtual Reality-based Simulation Prior to Lumbar Transforaminal Injections
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Sunmin Kim, Clinical Assistant Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: VRTF
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radiculopathy; virtual reality; Transforaminal epidural steroid injection; virtual simulator
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR simulation (Experimental): In this group, the practitioner will perform lumbar transforaminal epidural steroid injections after undergoing training using a 3D virtual simulator based on the patient's CT images.
  Interventions: Device: Virtual reality simulator
- Conventional (No Intervention): In this group, the patients will undergo lumbar transforaminal epidural steroid injections without the practitioner receiving any additional training.

INTERVENTIONS:
Device: Virtual reality simulator — This virtual reality simulator allows for the simulation of a lumbar transforaminal epidural steroid injection using the patient's 3D lumbar images.
  Arms: VR simulation

SUMMARY:
This study aims to evaluate the impact of pre-procedure training using a 3D simulator, based on lumbar CT images, on the success rate and efficiency of lumbar transforaminal steroid injections in patients who are expected to be difficult to treat. The training is provided to practitioners prior to performing the procedure on these patients.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of pre-procedure training using a 3D simulator, based on lumbar CT images, on the success rate and efficiency of lumbar transforaminal steroid injections in patients who are expected to be difficult to treat. The training is provided to practitioners prior to performing the procedure on these patients.

The lumbar transforaminal epidural steroid injection (TFESI) is a widely used non-surgical treatment for chronic lower back pain and sciatica. TFESI is effective in reducing inflammation and alleviating pain, but the procedure can be challenging due to anatomical structures and individual variations. In particular, when chronic degenerative changes in the lower back, such as reduced disc height, hypertrophy of the facet joints, foraminal stenosis, lateral recess hypertrophy, and the formation of osteophytes, complicate the needle insertion path or increase the likelihood of the needle contacting bone, a high level of skill and experience is required.

Recently, advancements in virtual reality (VR) technology have enabled highly realistic 3D simulations, which have spurred a growing body of research on VR-based simulations in healthcare. These simulations range from complex surgeries to disaster preparedness training in hospital settings. VR-based simulations offer an environment similar to real procedures, allowing practitioners to improve their skills and providing opportunities to rehearse complex or difficult cases in advance.

However, despite the growing interest in VR simulations across various fields, research on their application to precise procedures like TFESI remains scarce. To the best of our knowledge, no studies have utilized real patient imaging to create 3D models in a virtual environment for this purpose.

This study, against this background, aims to evaluate the impact of 3D virtual reality simulations using lumbar CT images of actual patients on the outcomes of transforaminal epidural steroid injections through a randomized controlled trial. The study will clarify how VR simulations can alleviate procedural difficulties and improve success rates and patient satisfaction compared to conventional image assessment methods. Moreover, it will contribute to establishing the foundation for incorporating VR-based simulations into standard protocols for complex procedures in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar lateral recess or foraminal stenosis who are scheduled to undergo lumbar transforaminal epidural steroid injection.
* Patients with lumbar CT images, where all four pain specialists in anesthesiology and pain medicine have determined that needle insertion through the transforaminal approach would be difficult.

Exclusion Criteria:

* Patients who have previously undergone transforaminal epidural steroid injections at this center.
* Patients with abnormal lumbar anatomical structures or a history of lumbar surgery.
* Patients who do not consent to participate in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Procedure time (seconds) | Immediately after the procedure
  The time taken to perform each procedure will be measured in seconds.
Number of fluoroscopic image shots | Immediately after the procedure
  The number of fluoroscopic image shots taken will be measured.

SECONDARY OUTCOMES:
Number of bone contacts | Immediately after the procedure
  The number of times the needle tip contacts the bone will be measured based on the practitioner's tactile feedback.
Patient satisfaction | Immediately after the procedure
  After the procedure, patient satisfaction will be assessed using a questionnaire consisting of four items, with responses measured on a 5-point Likert scale ranging from "strongly agree" to "strongly disagree."
Presence of vascular injection | Immediately after the procedure
  The procedure image will be analyzed to determine whether contrast dye was visualized in the blood vessels, confirming the presence or absence of intravascular injection.
Procedure success or failure | Immediately after the procedure
  The success or failure of the procedure, as determined by the practitioner, will be recorded.